CLINICAL TRIAL: NCT00805077
Title: Pulmonary Surgery and Protective Mechanical Ventilation
Acronym: VPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P070119
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Lung Neoplasms
Keywords: interoperative care; Tidal volume; Postoperative complications; Pneumonectomy; Lobectomy; Mechanical ventilation
MeSH Terms: conditions — Lung Neoplasms; Postoperative Complications | interventions — Respiration, Artificial; Tidal Volume

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): mechanical ventilation with low tidal volume (5 ml/kg of ideal body weight) plus PEEP
  Interventions: Procedure: mechanical ventilation
- 2 (Other): tidal volume of 10 ml/kg of ideal body weight without PEEP
  Interventions: Other: tidal volume

INTERVENTIONS:
Procedure: mechanical ventilation — mechanical ventilation with low tidal volume (5 ml/kg of ideal body weight) plus PEEP
  Arms: 1
Other: tidal volume — tidal volume of 10 ml/kg of ideal body weight without PEEP
  Arms: 2

SUMMARY:
The purpose of this trial is to evaluate the efficacy and the safety of lung protective ventilation during anesthesia in patients undergoing pneumonectomy or lobectomy for lung cancer.

DETAILED DESCRIPTION:
Extended description of the protocol could be provided by the URC-EST, SAINT ANTOINE HOSPITAL, University of Paris-VI and by principal investigator.

Pneumonectomy or lobectomy is associated with a high risk for postoperative complication. The benefit of lung protective ventilation with low tidal volume has been demonstrated in patients with acute respiratory distress syndrome (ARDS) and acute lung injury (ALI). Recent clinical studies have suggested that mechanical ventilation with low tidal volume may also profit in others setting. Lung protective ventilation during anaesthesia has been found to limit the inflammatory response in the lung and to decrease postoperative systemic inflammatory response. However, others trials did not found benefit of protective ventilation strategy during anaesthesia.

This study will be a randomized, controlled, doubled blind trial comparing two management ventilator strategies during anaesthesia for thoracotomy. Only patients undergoing pneumonectomy or lobectomy for lung primitive cancer will be included in this trial. During anesthesia, one group will receive mechanical ventilation with low tidal volume (5 ml/kg of ideal body weight) plus PEEP and the other will receive tidal volume of 10 ml/kg of ideal body weight without PEEP. After surgery, data concerning oxygen delivery, blood analysis, complications, cancer recurrence and death will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung cancer.
* Elective Pneumonectomy or lobectomy or bilobectomy
* Written informed consent

Exclusion Criteria:

* Patients undergoing surgical procedure other than pneumonectomy or lobectomy or bilobectomy
* Mesothelioma
* Liver cirrhosis
* Chronic renal failure
* Need for mechanical ventilation or non invasive ventilation (CPAP for obstructive sleep apnea syndrome for example) before surgery
* Emergency surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Major postoperative complications during the first 30 days after surgery | the first 30 days after surgery

SECONDARY OUTCOMES:
Minor postoperative complications during the first 30 days after surgery, length of stay in ICU and hospital, cancer recurrence, death | during the first 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Marret, MD, Principal Investigator — Hopital Tenon, Assistance Publique - Hopitaux de Paris
Locations (1):
- Departement d'Anesthesie Reanimation, Hopital Tenon, Paris, France

REFERENCES:
- [Derived] Marret E, Cinotti R, Berard L, Piriou V, Jobard J, Barrucand B, Radu D, Jaber S, Bonnet F; and the PPV study group. Protective ventilation during anaesthesia reduces major postoperative complications after lung cancer surgery: A double-blind randomised controlled trial. Eur J Anaesthesiol. 2018 Oct;35(10):727-735. doi: 10.1097/EJA.0000000000000804. PMID 29561278